CLINICAL TRIAL: NCT01439360
Title: An Efficacy Study of GSK Biologicals' Quadrivalent Influenza Vaccine GSK2321138A (FLU D-QIV) When Administered in Children
Brief Title: An Efficacy Study of GlaxoSmithKline (GSK) Biologicals' Candidate Influenza Vaccine GSK2321138A in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 115345; 2011-000758-41 (EudraCT Number)
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Influenza
Keywords: Vaccine; Seasonal Flu; Efficacy; Children
MeSH Terms: conditions — Influenza, Human | interventions — 13-valent pneumococcal vaccine; Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- D-QIV (Experimental): Subjects received 1 or 2 doses of candidate influenza Influsplit™ Tetra vaccine (GSK2321138A).
  Interventions: Biological: Quadrivalent seasonal influenza vaccine(Flu D-QIV) GSK2321138A
- Control (Active Comparator): In function of their age and D-QIV-vaccine status, subjects received Prevenar 13® or Havrix® Junior and possibly a varicella vaccine (Varilrix® or Varivax/ProVarivax ®).
  Interventions: Biological: Havrix Junior; Biological: Prevenar 13; Biological: Varivax/ProVarivax; Biological: Varilrix

INTERVENTIONS:
Biological: Quadrivalent seasonal influenza vaccine(Flu D-QIV) GSK2321138A — Intramuscular injection
  Arms: D-QIV
Biological: Havrix Junior — Intramuscular injection administered to subjects aged 12 months or older
  Arms: Control
Biological: Prevenar 13 — Intramuscular injection administered to subjects less than 12 months of age
  Arms: Control
Biological: Varivax/ProVarivax — Intramuscular injection administered to subjects more than 12 months of age
  Arms: Control
Biological: Varilrix — Subcutaneous injection administered to subjects more than 12 months of age
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the efficacy, immunogenicity and safety of GSK Biologicals' influenza candidate vaccine GSK2321138A when compared to non-influenza vaccine comparators in children 6 to 35 months of age. Recruitment will encompass at least 4 independent cohorts: a first cohort in the Northern Hemisphere (2011-2012), a second cohort in subtropical countries (2012), third cohort in the Northern Hemisphere (2012-2013) and a fourth cohort and additional independent cohorts possibly in NH countries (end 2013) and subtropical countries (beginning 2014).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/Legally Acceptable Representative (LARs) can and will comply with the requirements of the protocol.
* A male or female between, and including, 6 and 35 months of age at the time of first vaccination; children are eligible regardless of history of influenza vaccination.
* Written informed consent obtained from the parent(s) /LAR(s) of the subject.
* Subjects in stable health as determined by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Participation in a previous FLU-D-QIV-004 study (115345) cohort.
* Child in care.
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Prior receipt of any influenza vaccine within 6 months preceding the first dose of study vaccine, or planned use of such vaccines during the study period.
* Children with underlying illness who are at risk of complications of influenza and for whom yearly (seasonal) influenza vaccination is recommended in their respective country.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (including HIV), based on medical history and physical examination.
* Chronic administration of immunosuppressants or other immune modifying drugs within six months prior to the first vaccine dose. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/ or any blood products within 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines, non-influenza vaccine comparators and latex; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous vaccination.
* Any contraindication to intramuscular injection.
* Acute disease and/or fever at the time of enrolment.
* Any other condition which, in the opinion of the Investigator, prevents the subject from participating in the study.
* Additional criteria for children ≥ 12 months of age:

  * Prior receipt of any licensed varicella vaccine* or any licensed hepatitis A vaccine or planned use of these vaccines during the study period. Other routine registered childhood vaccinations are permitted.

    * For countries with varicella vaccine administered as 2-dose schedule, prior receipt of a single dose of a varicella vaccine is allowed if administered at least 2 weeks before the first study vaccination.
  * Any history of hepatitis A or varicella diseases.
* Additional criteria for children 6 - 11 months of age in countries without universal mass vaccination recommendation for pneumococcal vaccine:

  * Prior receipt of any pneumococcal conjugated vaccine or planned use of this vaccine during the study period. Other routine registered childhood vaccinations are permitted.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12046 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (87):
- GSK Investigational Site, Dhaka, Bangladesh
- Belgium (6):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Mechelen
  - GSK Investigational Site, Namur
  - GSK Investigational Site, Roeselaere
  - GSK Investigational Site, Turnhout
- Czechia (11):
  - GSK Investigational Site, Děčín
  - GSK Investigational Site, Humpolec
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Lipník nad Bečvou
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Odolena Voda
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Tábor
- Dominican Republic (2):
  - GSK Investigational Site, Santo Domingo
  - GSK Investigational Site, Santo Domingo, Distrito Nacional
- Honduras (2):
  - GSK Investigational Site, San Pedro Sula
  - GSK Investigational Site, Tegucigalpa
- India (2):
  - GSK Investigational Site, Faridabad
  - GSK Investigational Site, Pune
- GSK Investigational Site, Beirut, Lebanon
- Philippines (5):
  - GSK Investigational Site, City of Muntinlupa
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Metro Manila
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, Sampaloc, Manila
- Poland (17):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Oborniki
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wola
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Łęczna
- Spain (15):
  - GSK Investigational Site, Antequera/Málaga
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Blanes (Girona)
  - GSK Investigational Site, Boadilla del Monte
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Quart de Poblet, Valencia
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Torrelodones (Madrid)
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vic/ Barcelona
  - GSK Investigational Site, Xativa/Valencia
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Bursa
  - GSK Investigational Site, Eskişehir
  - GSK Investigational Site, Istanbul
- United Kingdom (20):
  - GSK Investigational Site, St Austell, Cornwall
  - GSK Investigational Site, Southampton, Hampshire
  - GSK Investigational Site, Axbridge, Somerset
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Yeovil, Somerset
  - GSK Investigational Site, Atherstone, Warwickshire
  - GSK Investigational Site, Coventry, Warwickshire
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Bolton, Nr Manchester
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Co Antrim
  - GSK Investigational Site, Crumpsall, Manchester
  - GSK Investigational Site, Exeter
  - GSK Investigational Site, Gloucester
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Taunton, Somerset
  - GSK Investigational Site, Westminster Bridge Road

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Danier J, Callegaro A, Soni J, Carmona A, Kosalaraska P, Rivera L, Friel D, Pu W, Vantomme V, Dbaibo G, Innis BL, Schuind A, Zaman K, Wilson J. Association Between Hemagglutination Inhibition Antibody Titers and Protection Against Reverse-Transcription Polymerase Chain Reaction-Confirmed Influenza Illness in Children 6-35 Months of Age: Statistical Evaluation of a Correlate of Protection. Open Forum Infect Dis. 2021 Sep 25;9(2):ofab477. doi: 10.1093/ofid/ofab477. eCollection 2022 Feb. PMID 35083365
- [Derived] Dbaibo G, Amanullah A, Claeys C, Izu A, Jain VK, Kosalaraksa P, Rivera L, Soni J, Yanni E, Zaman K, Acosta B, Ariza M, Arroba Basanta ML, Bavdekar A, Carmona A, Cousin L, Danier J, Diaz A, Diez-Domingo J, Dinleyici EC, Faust SN, Garcia-Sicilia J, Gomez-Go GD, Gonzales MLA, Hacimustafaoglu M, Hughes SM, Jackowska T, Kant S, Lucero M, Mares Bermudez J, Martinon-Torres F, Montellano M, Prymula R, Puthanakit T, Ruzkova R, Sadowska-Krawczenko I, Szymanski H, Ulied A, Woo W, Schuind A, Innis BL; Flu4VEC Study Group. Quadrivalent Influenza Vaccine Prevents Illness and Reduces Healthcare Utilization Across Diverse Geographic Regions During Five Influenza Seasons: A Randomized Clinical Trial. Pediatr Infect Dis J. 2020 Jan;39(1):e1-e10. doi: 10.1097/INF.0000000000002504. PMID 31725115
- [Derived] Danier J, Rivera L, Claeys C, Dbaibo G, Jain VK, Kosalaraksa P, Woo W, Yanni E, Zaman K, Acosta B, Amanullah A, Ariza M, Luisa Arroba Basanta M, Bavdekar A, Carmona A, Cousin L, Diaz A, Diez-Domingo J, Cagri Dinleyici E, Faust SN, Garcia-Sicilia J, Gomez-Go GD, Antionette Gonzales L, Hacimustafaoglu M, Hughes SM, Izu A, Jackowska T, Kant S, Lucero M, Mares Bermudez J, Martinon-Torres F, Montellano M, Prymula R, Puthanakit T, Ruzkova R, Sadowska-Krawczenko I, Soni J, Szymanski H, Ulied A, Schuind A, Innis BL; Flu4VEC Study Group. Clinical Presentation of Influenza in Children 6 to 35 Months of Age: Findings From a Randomized Clinical Trial of Inactivated Quadrivalent Influenza Vaccine. Pediatr Infect Dis J. 2019 Aug;38(8):866-872. doi: 10.1097/INF.0000000000002387. PMID 31306399
- [Derived] Claeys C, Chandrasekaran V, Garcia-Sicilia J, Prymula R, Diez-Domingo J, Brzostek J, Mares-Bermudez J, Martinon-Torres F, Pollard AJ, Ruzkova R, Carmona Martinez A, Ulied A, Miranda Valdivieso M, Faust SN, Snape MD, Friel D, Ollinger T, Soni J, Schuind A, Li P, Innis BL, Jain VK. Anamnestic Immune Response and Safety of an Inactivated Quadrivalent Influenza Vaccine in Primed Versus Vaccine-Naive Children. Pediatr Infect Dis J. 2019 Feb;38(2):203-210. doi: 10.1097/INF.0000000000002217. PMID 30325891
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 12046 enrolled subjects, 21 subjects were excluded from all statistical analyses due to an invalid informed consent form (ICF) and 7 subjects did not receive any study vaccine despite being allocated a subject number, hence only 12018 subjects started this study.
Groups:
- Control: In function of their age and Influsplit™ Tetra (D-QIV) vaccine status, subjects received Prevenar 13® or Havrix® Junior and possibly a varicella vaccine (Varilrix® or Varivax/ProVarivax ®).
Period: Overall Study
Arm/Group | D-QIV | Control
Started | 6006 | 6012
Completed | 5808 | 5804
Not Completed | 198 | 208
Not completed — Adverse Event | 4 | 16
Not completed — Lost to Follow-up | 43 | 58
Not completed — Others | 10 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 140 | 129

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-QIV | Control | Total
Number analyzed (Participants) | 6006 | 6012 | 12018
Age, Continuous [Mean (Standard Deviation); unit: Months] | 21.9 (8.0) | 21.8 (8.0) | 21.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2933 | 2925 | 5858
  Male | 3073 | 3087 | 6160
Race/Ethnicity, Customized [Number; unit: Participants]
  African Heritage / African American | 24 | 20 | 44
  Asian - Central/South Asian Heritage | 1062 | 1053 | 2115
  Asian - East Asian Heritage | 2 | 0 | 2
  Asian - Japanese Heritage | 2 | 0 | 2
  Asian - South East Asian Heritage | 1661 | 1666 | 3327
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Other | 1639 | 1642 | 3281
  White - Arabic / North African Heritage | 142 | 149 | 291
  White - Caucasian / European Heritage | 1471 | 1482 | 2953

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Moderate to Severe RT-PCR Confirmed Influenza.
Description: Attack rate (AR) was defined as the number/percentage of subjects with at least 1 RT-PCR confirmed influenza event.
Time Frame: During the surveillance period (approximately 6 to 8 months)
Population: The ATP cohort for efficacy - Time to event included all eligible subjects who received study vaccine(s) according to their random assignment, for whom vaccine administration site was known, who had a swab collected during the window (0-7 days) of episode onset and who would be censored but not eliminated based on protocol criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 5707 | 5697
Participants | 90 | 242
Statistical Analysis 1: Comparison: D-QIV vs Control; The efficacy of the D-QIV vaccine would be demonstrated if the LL of the two-sided 97.5% CI for vaccine efficacy (VE) is above (>) 25%; Test type: Superiority or Other; Regression, Cox; Adjusted for age category and stratified for cohort; Vaccine efficacy (VE) = 63.2, 97.5% CI 2-sided [51.8 to 72.3] — VE was defined as the hazard ratio of cases of influenza A and or B disease in subjects receiving D-QIV vaccine in contrast with subjects receiving non-influenza vaccine control subtracted from 1

2. Primary Outcome: Number of Subjects With RT-PCR Confirmed Influenza of Any Severity.
Description: Attack rate (AR) was defined as the number/percentage of subjects with at least 1 RT-PCR confirmed influenza event.
Time Frame: During the surveillance period (approximately 6 to 8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 5707 | 5697
Participants | 344 | 662
Statistical Analysis 1: Comparison: D-QIV vs Control; The efficacy of the D-QIV vaccine would be demonstrated if the LL of the two-sided 97.5% CI for VE is above 15%; Test type: Superiority or Other; Regression, Cox; Adjusted for age category and stratified for cohort; Vaccine efficacy (VE) = 49.8, 97.5% CI 2-sided [41.8 to 56.8] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Subjects With First Occurrence of Lower Respiratory Illness (LRI) With RT-PCR Confirmed Influenza.
Description: Attack rate (AR) was defined as the number/percentage of subjects with at least 1 RT-PCR confirmed influenza event.
Time Frame: At any time starting 7 days before the onset of LRI and ending 7 days after end of LRI during the surveillance period (approximately 6 to 8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 5707 | 5697
Participants | 28 | 61

4. Secondary Outcome: Number of Subjects With First Occurrence of Culture-confirmed Moderate to Severe Influenza A and/or B Disease Due to Antigenically-matching Influenza Strains.
Description: Attack rate (AR) was defined as the number/percentage of subjects with at least 1 RT-PCR confirmed influenza event.
Time Frame: During the surveillance period (approximately 6 to 8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 5707 | 5697
Participants | 20 | 88

5. Secondary Outcome: Number of Subjects With First Occurrence of Culture-confirmed Influenza A and/or B Disease of Any Severity Due to Antigenically-matching Influenza Strains
Description: Attack rate (AR) was defined as the number/percentage of subjects with at least 1 RT-PCR confirmed influenza event.
Time Frame: During the surveillance period (approximately 6 to 8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 5707 | 5697
Participants | 88 | 216

6. Secondary Outcome: Number of Subjects With First Occurrence of Culture-confirmed Moderate to Severe Influenza A and/or B Disease Due to Any Seasonal Influenza Strain.
Description: Attack rate (AR) was defined as the number/percentage of subjects with at least 1 RT-PCR confirmed influenza event.
Time Frame: During the surveillance period (approximately 6 to 8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 5707 | 5697
Participants | 79 | 216

7. Secondary Outcome: Number of Subjects With First Occurrence of Culture-confirmed Influenza A and/or B Disease of Any Severity Due to Any Seasonal Influenza Strain.
Description: Attack rate (AR) was defined as the number/percentage of subjects with at least 1 RT-PCR confirmed influenza event.
Time Frame: During the surveillance period (approximately 6 to 8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 5707 | 5697
Participants | 303 | 602

8. Secondary Outcome: Number of Subjects With First Occurrence of Acute Otitis Media (AOM) With RT-PCR Confirmed Influenza A and/or B Infection Due to Any Seasonal Influenza Strain.
Description: Attack rate (AR) was defined as the number/percentage of subjects with at least 1 RT-PCR confirmed influenza event.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 5707 | 5697
Participants | 12 | 28

9. Secondary Outcome: Number of Subjects With First Occurrence of RT-PCR Confirmed Severe Influenza A and/or B Due to Any Seasonal Influenza Strain.
Description: Attack rate (AR) was defined as the number/percentage of subjects with at least 1 RT-PCR confirmed influenza event.
Time Frame: During the surveillance period (approximately 6 to 8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 5707 | 5697
Participants | 2 | 3

10. Secondary Outcome: Humoral Immune Response in Terms of Haemagglutination-inhibition (HI) Antibody Titres Against Each of Four Vaccine Strains Contained in the D-QIV (in Immuno Subcohort of Subjects Only)
Description: Titers were expressed as geometric mean antibody titers (GMTs). The vaccine strains assessed were A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Brisbane/3/2007 (Yamagata).
  PRE= Pre-vaccination at Day 0; POST = Post-vaccination 1 at Day 28 for primed subjects or post-vaccination 2 at Day 56 for unprimed subjects
Time Frame: At Days 0 and 28/56
Population: The ATP cohort for immunogenicity included all evaluable subjects for whom data concerning immunogenicity outcome measures were available. These included subjects for whom assay results were available for antibodies against at least one study vaccine strain after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 753 | 579
Titers
  H1N1, PRE: number analyzed (Participants) | 744 | 567
  H1N1, PRE | 11.9 [10.6 to 13.2] | 11.9 [10.5 to 13.5]
  H1N1, POST: number analyzed (Participants) | 752 | 578
  H1N1, POST | 165.3 [148.6 to 183.8] | 12.6 [11.1 to 14.3]
  H3N2, PRE: number analyzed (Participants) | 746 | 568
  H3N2, PRE | 14.8 [13.2 to 16.5] | 13.4 [11.8 to 15.2]
  H3N2, POST: number analyzed (Participants) | 753 | 578
  H3N2, POST | 132.1 [119.1 to 146.5] | 14.7 [12.9 to 16.7]
  Victoria, PRE: number analyzed (Participants) | 745 | 567
  Victoria, PRE | 10.0 [9.1 to 11.0] | 9.2 [8.3 to 10.1]
  Victoria, POST: number analyzed (Participants) | 750 | 579
  Victoria, POST | 92.6 [82.3 to 104.1] | 9.2 [8.4 to 10.1]
  Yamagata, PRE: number analyzed (Participants) | 745 | 568
  Yamagata, PRE | 7.3 [6.8 to 7.8] | 7.3 [6.8 to 7.9]
  Yamagata, POST | 121.4 [110.1 to 133.8] | 7.6 [7.0 to 8.3]

11. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies Against Each of the 4 Influenza Strains Contained in the D-QIV Vaccine (in Immuno Subcohort of Subjects Only)
Description: A seropositive subject was a subject whose HI antibody titer was greater than or equal to the assay cut-off value of 1:10. The vaccine strains assessed were A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Brisbane/3/2007 (Yamagata).
  PRE= Pre-vaccination at Day 0; POST = Post-vaccination 1 at Day 28 for primed subjects or post-vaccination 2 at Day 56 for unprimed subjects.
Time Frame: At Day 0 and Day 28/56
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 753 | 579
Participants
  H1N1, PRE | 200 | 152
  H1N1, POST | 728 | 170
  H3N2, PRE | 266 | 187
  H3N2, POST | 740 | 210
  Victoria, PRE | 205 | 138
  Victoria, POST | 701 | 147
  Yamagata, PRE | 134 | 93
  Yamagata, POST | 719 | 108

12. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against Each of the 4 Influenza Strains Contained in the D-QIV Vaccine (in Immuno Subcohort of Subjects Only)
Description: Seroconversion rate (SCR) was defined as the number of subjects who have either a pre-vaccination reciprocal HI titer < 1:10 and a post-vaccination reciprocal titer ≥ 1:40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4 fold increase in post vaccination reciprocal titer against the vaccine virus.
  PRE= Pre-vaccination at Day 0; POST = Post-vaccination 1 at Day 28 for primed subjects or post-vaccination 2 at Day 56 for unprimed subjects
Time Frame: At Day 28/56 (POST)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 746 | 568
Participants
  H1N1 | 596 | 20
  H3N2 | 513 | 24
  Victoria | 514 | 5
  Yamagata | 605 | 13

13. Secondary Outcome: Mean Geometric Increase (MGI) for HI Antibody Titer Against Each of the 4 Vaccine Influenza Strains Contained in the D-QIV Vaccine (in Immuno Subcohort of Subjects Only).
Description: MGI also known as the seroconversion factor [SCF] was defined as the fold increase in serum HI GMTs post vaccination compared to pre-vaccination (Day 0). The vaccine strains assessed were A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Brisbane/3/2007 (Yamagata).
  POST = Post-vaccination 1 at Day 28 for primed subjects or post-vaccination 2 at Day 56 for unprimed subjects.
Time Frame: At Day 28/56 (POST)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 746 | 568
Fold change
  H1N1 | 14 [12.8 to 15.3] | 1.1 [1.0 to 1.1]
  H3N2 | 9.0 [8.2 to 9.8] | 1.1 [1.0 to 1.2]
  Victoria | 9.3 [8.6 to 10.2] | 1.0 [1.0 to 1.1]
  Yamagata | 16.7 [15.2 to 18.3] | 1.1 [1.0 to 1.1]

14. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies Against Each of the 4 Influenza Strains Contained in the D-QIV Vaccine (in Immuno Subcohort of Subjects Only)
Description: Seroprotection rate (SPR) was defined as the number of subjects with H1N1 reciprocal HI titers ≥ 1:40 against the tested vaccine virus.The vaccine strains assessed were A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Brisbane/3/2007 (Yamagata).
  PRE= Pre-vaccination at Day 0; POST = Post-vaccination 1 at Day 28 for primed subjects or post-vaccination 2 at Day 56 for unprimed subjects
Time Frame: At Day 0 and Day 28/56
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 753 | 579
Participants
  H1N1, PRE | 182 | 134
  H1N1, POST | 640 | 146
  H3N2, PRE | 238 | 159
  H3N2, POST | 612 | 175
  Victoria, PRE | 143 | 103
  Victoria, POST | 539 | 101
  Yamagata, PRE | 73 | 59
  Yamagata, POST | 638 | 64

15. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as pain that resulted crying when limb was moved/ spontaneously painful. Grade 3 redness and swelling was greater than 50 millimeters (mm) i.e. >50mm.
Time Frame: During the 7-day post-vaccination period (Days 0-6 for Dose 1, Days 28-34 for Dose 2)
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented. The analysis of solicited symptoms based on the Total Vaccinated cohort included only subjects/doses with documented safety data (i.e. symptom screen/sheet completed).
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 5907 | 5901
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 5899 | 5896
  Any Pain, Dose 1 | 1015 | 1047
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 5899 | 5896
  Grade 3 Pain, Dose 1 | 23 | 30
  Any Redness, Dose 1: number analyzed (Participants) | 5899 | 5896
  Any Redness, Dose 1 | 775 | 831
  Grade 3 Redness, Pain, Dose 1: number analyzed (Participants) | 5899 | 5896
  Grade 3 Redness, Pain, Dose 1 | 1 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 5899 | 5896
  Any Swelling, Dose 1 | 467 | 518
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 5899 | 5896
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 5757 | 5766
  Any Pain, Dose 2 | 808 | 820
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 5757 | 5766
  Grade 3 Pain, Dose 2 | 21 | 21
  Any Redness, Dose 2: number analyzed (Participants) | 5757 | 5766
  Any Redness, Dose 2 | 587 | 631
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 5757 | 5766
  Grade 3 Redness, Dose 2 | 2 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 5757 | 5766
  Any Swelling, Dose 2 | 375 | 409
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 5757 | 5766
  Grade 3 Swelling, Dose 2 | 2 | 3
  Any Pain, Across doses | 1350 | 1375
  Grade 3 Pain, Across doses | 42 | 48
  Any Redness, Across doses | 980 | 1091
  Grade 3 Redness, Across doses | 3 | 0
  Any Swelling, Across doses | 665 | 742
  Grade 3 Swelling, Across doses | 2 | 3

16. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were Drowsiness, Irritability/fussiness, Loss of appetite and Temperature (Axillary). Any was defined as any general symptom reported irrespective of intensity or relationship to vaccination. Grade 3 was defined as symptoms that prevented normal activity. Related was defined as general symptom assessed by the investigator to have a causal relationship to vaccination.
Time Frame: During the 7-day post-vaccination period (Days 0-6 for Dose 1, Days 28-34 for Dose 2)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 5908 | 5901
Participants
  Any Drowsiness, Dose 1: number analyzed (Participants) | 5898 | 5896
  Any Drowsiness, Dose 1 | 739 | 829
  Grade 3 Drowsiness, Dose 1: number analyzed (Participants) | 5898 | 5896
  Grade 3 Drowsiness, Dose 1 | 39 | 52
  Related Drowsiness, Dose 1: number analyzed (Participants) | 5898 | 5896
  Related Drowsiness, Dose 1 | 490 | 535
  Any Irritability, Dose 1: number analyzed (Participants) | 5898 | 5896
  Any Irritability, Dose 1 | 955 | 1029
  Grade 3 Irritability, Dose 1: number analyzed (Participants) | 5898 | 5896
  Grade 3 Irritability, Dose 1 | 42 | 62
  Related Irritability, Dose 1: number analyzed (Participants) | 5898 | 5896
  Related Irritability, Dose 1 | 617 | 669
  Any Loss of appetite, Dose 1: number analyzed (Participants) | 5898 | 5896
  Any Loss of appetite, Dose 1 | 847 | 872
  Grade 3 Loss of appetite, Dose 1: number analyzed (Participants) | 5898 | 5896
  Grade 3 Loss of appetite, Dose 1 | 68 | 60
  Related Loss of appetite, Dose 1: number analyzed (Participants) | 5898 | 5896
  Related Loss of appetite, Dose 1 | 541 | 523
  Any Fever, Dose 1: number analyzed (Participants) | 5898 | 5896
  Any Fever, Dose 1 | 372 | 425
  Grade 3 Fever, Dose 1: number analyzed (Participants) | 5898 | 5896
  Grade 3 Fever, Dose 1 | 78 | 76
  Related Fever, Dose 1: number analyzed (Participants) | 5898 | 5896
  Related Fever, Dose 1 | 243 | 287
  Any Drowsiness, Dose 2: number analyzed (Participants) | 5755 | 5762
  Any Drowsiness, Dose 2 | 519 | 558
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 5755 | 5762
  Grade 3 Drowsiness, Dose 2 | 25 | 24
  Related Drowsiness, Dose 2: number analyzed (Participants) | 5755 | 5762
  Related Drowsiness, Dose 2 | 324 | 361
  Any Irritability, Dose 2: number analyzed (Participants) | 5755 | 5762
  Any Irritability, Dose 2 | 777 | 777
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 5755 | 5762
  Grade 3 Irritability, Dose 2 | 36 | 52
  Related Irritability, Dose 2: number analyzed (Participants) | 5755 | 5762
  Related Irritability, Dose 2 | 488 | 495
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 5755 | 5762
  Any Loss of appetite, Dose 2 | 652 | 681
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 5755 | 5762
  Grade 3 Loss of appetite, Dose 2 | 47 | 44
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 5755 | 5762
  Related Loss of appetite, Dose 2 | 378 | 413
  Any Fever, Dose 2: number analyzed (Participants) | 5755 | 5762
  Any Fever, Dose 2 | 336 | 363
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 5755 | 5762
  Grade 3 Fever, Dose 2 | 65 | 70
  Related Fever, Dose 2: number analyzed (Participants) | 5755 | 5762
  Related Fever, Dose 2 | 195 | 215
  Any Drowsiness, Across Doses | 1024 | 1129
  Grade 3 Drowsiness, Across Doses | 61 | 73
  Related Drowsiness, Across Doses | 673 | 738
  Any Irritability, Across Doses | 1383 | 1427
  Grade 3 Irritability, Across Doses | 77 | 107
  Related Irritability, Across Doses | 905 | 940
  Any Loss of appetite, Across Doses | 1227 | 1288
  Grade3 Loss of appetite,Across Doses | 111 | 97
  Related Loss of appetite,AcrossDoses | 774 | 809
  Any Fever, Across Doses | 659 | 732
  Grade 3 Fever, Across Doses | 137 | 141
  Related Fever, Across Doses | 413 | 476

17. Secondary Outcome: Duration of Solicited Local Symptoms
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: During the 7-day post-vaccination period (Days 0-6 for Dose 1, Days 28-34 for Dose 2)
Population: as for outcome 15
Measure: Median (Full Range); unit: Days
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 1015 | 1047
Days
  Pain, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Pain, Dose 2: number analyzed (Participants) | 808 | 820
  Pain, Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Redness, Dose 1: number analyzed (Participants) | 775 | 831
  Redness, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Redness, Dose 2: number analyzed (Participants) | 587 | 631
  Redness, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Swelling, Dose 1: number analyzed (Participants) | 467 | 518
  Swelling, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Swelling, Dose 2: number analyzed (Participants) | 375 | 409
  Swelling, Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]

18. Secondary Outcome: Duration of Solicited General Symptoms
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: During the 7-day post-vaccination period (Days 0-6 for Dose 1, Days 28-34 for Dose 2)
Population: as for outcome 15
Measure: Median (Full Range); unit: Days
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 955 | 1029
Days
  Drowsiness, Dose 1: number analyzed (Participants) | 739 | 829
  Drowsiness, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Drowsiness, Dose 2: number analyzed (Participants) | 519 | 558
  Drowsiness, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Irritability, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Irritability, Dose 2: number analyzed (Participants) | 777 | 777
  Irritability, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Loss of appetite, Dose 1: number analyzed (Participants) | 847 | 872
  Loss of appetite, Dose 1 | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0]
  Loss of appetite, Dose 2: number analyzed (Participants) | 652 | 681
  Loss of appetite, Dose 2 | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 4.0]
  Fever, Dose 1: number analyzed (Participants) | 390 | 438
  Fever, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Fever, Dose 2: number analyzed (Participants) | 347 | 372
  Fever, Dose 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]

19. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the 28-day (Days 0-27) post-vaccination period
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 6006 | 6012
Participants
  Any unsolicited AEs | 2640 | 2679
  Grade 3 unsolicited AEs | 160 | 149
  Related unsolicited AEs | 106 | 116

20. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related AEs With Medically Attended Visits (MAVs)
Description: MAVs were defined as AEs with a medically-attended visit i.e. prompting emergency room (ER) visits, hospitalizations or physician visits and that were not routine visits for physical examination or vaccination. Any MAV was defined as at least one MAV experienced. Grade 3 was defined as MAVs that prevented normal activities and related was defined as MAVs assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the entire study period (approximately 6- 8 months per subject)
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 6006 | 6012
Participants
  Any MAVs | 3885 | 3988
  Grade 3 MAVs | 200 | 211
  Related MAVs | 57 | 58

21. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Potential Immune-mediated Diseases (pIMDs).
Description: pIMDs are a subset of adverse events (AEs) that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. Grade 3 = pIMDs that prevented normal activities. Related = symptom assed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (approximately 6- 8 months per subject)
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 6006 | 6012
Participants
  Any pIMDs | 5 | 0
  Grade 3 pIMDs | 3 | 0
  Related pIMDs | 3 | 0

22. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (approximately 6- 8 months per subject)
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-QIV | Control
Number analyzed (Participants) | 6006 | 6012
Participants
  Any SAEs | 217 | 201
  Related SAEs | 6 | 2
  Fatal SAEs | 1 | 3
  Related fatal SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms were assessed during the 7-day post-vaccination period (Days 0-6 for Dose 1, Days 28-34 for Dose 2); unsolicited AEs were assessed during the 28-day (Days 0-27) post-vaccination period; SAEs were reported during the entire study period (approximately 6- 8 months per subject)
Arm/Group | D-QIV | Control
Serious Adverse Events (participants affected / at risk) | 217/6006 | 201/6012
Other Adverse Events (participants affected / at risk) | 3427/6006 | 3501/6012
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-QIV (N=6006) | Control (N=6012)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypoplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 9 (9)
Gastritis (Gastrointestinal disorders) | 2 (3) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Drowning (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 4 (4)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Amoebiasis (Infections and infestations) | 3 (3) | 3 (3)
Amoebic dysentery (Infections and infestations) | 8 (8) | 3 (3)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Ascariasis (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 7 (7) | 6 (7)
Bronchitis (Infections and infestations) | 11 (12) | 9 (9)
Chest wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Chikungunya virus infection (Infections and infestations) | 0 (0) | 1 (1)
Cholera (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 1 (1)
Dengue fever (Infections and infestations) | 2 (2) | 10 (10)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 2 (2)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 27 (27) | 19 (20)
Gastroenteritis norovirus (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 5 (6) | 8 (8)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 2 (2)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 1 (1)
Hepatitis a (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Laryngitis (Infections and infestations) | 4 (4) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 6 (6) | 3 (3)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Mycoplasma infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Otitis media (Infections and infestations) | 4 (4) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 2 (2)
Parasitic gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 5 (5)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 56 (60) | 66 (71)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia measles (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 2 (2)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Typhoid fever (Infections and infestations) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (4)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Viral rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Viral sepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood electrolytes abnormal (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 8 (9) | 7 (7)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 13 (14) | 16 (16)
Seizure (Nervous system disorders) | 3 (3) | 2 (2)
Seizure anoxic (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 8 (8)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-QIV (N=6006) | Control (N=6012)
Decreased appetite (Metabolism and nutrition disorders) | 1230 (1504) | 1293 (1561)
Erythema (Skin and subcutaneous tissue disorders) | 983 (1365) | 1094 (1467)
Irritability (Psychiatric disorders) | 1385 (1734) | 1428 (1808)
Nasopharyngitis (Infections and infestations) | 871 (1050) | 943 (1111)
Pain (General disorders) | 1351 (1824) | 1376 (1868)
Pyrexia (General disorders) | 866 (954) | 949 (1042)
Somnolence (Nervous system disorders) | 1025 (1259) | 1129 (1388)
Swelling (General disorders) | 665 (842) | 743 (928)
Upper respiratory tract infection (Infections and infestations) | 522 (629) | 516 (609)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.